CLINICAL TRIAL: NCT01986387
Title: Virtual Peer-to-Peer (VP2P) Support Mentoring for Adolescents With Chronic Pain: A Feasibility Pilot Randomized Controlled Trial
Brief Title: Virtual Peer-to-Peer (VP2P) Support Mentoring for Chronic Pain: A Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Jennifer Stinson, Principal Investigator, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1000036188
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Chronic Pain
Keywords: adolescent; Skype; peer mentorship; internet self-management
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual Peer-to-Peer Support Mentoring (Experimental): In addition to standard medical care, adolescents in the experimental group will receive the VP2P support program, a manualized peer-mentorship program that will provide modeling and reinforcement by peers (young adults with chronic pain aged 16-25 years who have learned to function successfully with their chronic pain to the mentored participants).
  Interventions: Behavioral: Virtual Peer-to-Peer Support Mentoring
- Waitlist Control (No Intervention): The control group will receive usual care but without the mentorship intervention. They will be offered the VP2P support program after completion of outcome measures (T1 - to be completed online prior to randomization; T2 - at program completion).

INTERVENTIONS:
Behavioral: Virtual Peer-to-Peer Support Mentoring — The mentorship program will encourage mentored participants to develop and engage in self-management and transition skills and support their practice of these skills. The mentors will present information to mentored participants in a monitored virtual interaction using Skype for 8 weeks (10 total Skype sessions of 30-60 minutes each) to encourage participation in skill building tailored to their needs. All mentors will complete a paid 2.5 day training course and will be supported throughout the duration of the study (consultations with research staff to deal with unforeseen concerns). Mentored participants will complete online outcome measures prior to randomization (T1) and upon study completion (T2).
  Arms: Virtual Peer-to-Peer Support Mentoring

SUMMARY:
Study Hypothesis: A virtual peer-to-peer support intervention will improve health outcomes and quality of life in adolescents with chronic pain.

DETAILED DESCRIPTION:
The aim of this project is to develop and examine the impact of a virtual peer support program on health outcomes and quality of life of adolescents with chronic pain using a waitlist randomized controlled trial. In addition to standard medical care, adolescents in the experimental group will receive a manualized peer mentorship program that will provide modeling and reinforcement by trained young adults aged 16-25 years who have learned to function successfully with their pain. Mentoring sessions consist of 10 sessions of 30-45 minute Skype calls over 8 weeks. Feasibility of the program will be measured in addition to quality of life, physical and emotional symptoms, pain coping, self-efficacy, social support, and self-management skills.

ELIGIBILITY:
Inclusion Criteria:

* males and females 12-18 years old
* diagnosed chronic pain condition (e.g., neuropathic pain, Complex Regional Pain Syndrome, chronic musculoskeletal pain, chronic daily headache, chronic widespread pain)
* able to speak and read English
* access to Internet connection, computer capable of using free Skype software
* willing and able to complete online measures.

Exclusion Criteria:

* significant cognitive impairments
* major co-morbid illnesses (i.e., psychiatric conditions) likely to influence HRQL assessment
* participating in peer support or self-management interventions (e.g., WebMap).

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2015-05 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Feasibility | 2 months
  1. Accrual and Dropout Rates - recruitment and withdrawal rates will be calculated that the end of the study.
  2. Compliance (Level of Engagement) - rates of completion of weekly calls and online outcome measures will be calculated that the end of the study - defined as 100% when the participant completes 10 calls over 8 weeks with all online measures completed.
  3. Adolescents' Perception of Chronic Pain VP2P Program - the acceptability of and satisfaction with the Chronic Pain VP2P support program as measured through semi-structured phone interviews with mentees and focus groups with mentors
  4. Estimates of Intervention Effects (e.g., effect sizes, variance measures/standard deviation) on health outcomes to inform the calculation of an appropriate sample size for the future definitive multi-centred randomized controlled trial (RCT)

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQL) | Baseline, 2 months
  HRQL will be measured by using the 61-item Bath Adolescent Pain Questionnaire, which assesses the impact of chronic pain in adolescence in terms of physical, psychological and social functioning.
Emotional Symptoms | Baseline, 2 months
  Anxiety and depression will each be assessed using two, separate 8-item Patient Reported Outcomes Measurement Information System (PROMIS) scales.
Pain Coping | Baseline, 2 months
  Pain coping will be measured using the 18-item Pain Coping Questionnaire, which is an internationally used measure of pain coping strategies in the pediatric population.
Self-Efficacy | Baseline, 2 months
  Self-efficacy will be measured using a 10-item Pain Self-Efficacy Questionnaire (PSEQ) that assesses the confidence people have in performing activities while in pain.
Social Support | Baseline, 2 months
  Social support will be measured with the 12-item Multidimensional Scale of Perceived Social Support questionnaire that explores the impact that family, friends and significant others as social support.
Disability | Baseline, 2 months
  Disability will be measured using the 15-item Functional Disability Inventory, which assesses physical functioning and disability in youth with chronic pain.
Self-Management | Baseline, 2 months
  Self-management was measured using Self-Management Skills Assessment Guide, which was developed by Alberta Children's Hospital and consists of 21 items assessing adolescents' awareness of their health condition and ability to make decisions relevant to their health care needs (cite).
Pain | Baseline, 2 months
  Pain will be measured using the Brief Pain Inventory - Short Form (BPISF). The 9-item measure assesses the severity of pain and its impact on daily functions.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Stinson, RN,PhD,CPNP, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Result] Ahola Kohut S, Stinson JN, Ruskin D, Forgeron P, Harris L, van Wyk M, Luca S, Campbell F. iPeer2Peer program: a pilot feasibility study in adolescents with chronic pain. Pain. 2016 May;157(5):1146-1155. doi: 10.1097/j.pain.0000000000000496. PMID 26808145
- [Result] Ahola Kohut S, Stinson J, Forgeron P, Luca S, Harris L. Been There, Done That: The Experience of Acting as a Young Adult Mentor to Adolescents Living With Chronic Illness. J Pediatr Psychol. 2017 Oct 1;42(9):962-969. doi: 10.1093/jpepsy/jsx062. PMID 28340203
- [Result] Ahola Kohut S, Stinson J, Forgeron P, van Wyk M, Harris L, Luca S. A qualitative content analysis of peer mentoring video calls in adolescents with chronic illness. J Health Psychol. 2018 May;23(6):788-799. doi: 10.1177/1359105316669877. Epub 2016 Sep 28. PMID 27682341